CLINICAL TRIAL: NCT01044550
Title: Laparoscopy (to Detect Occult Diaphragm Injury) Versus Clinical and Radiological Follow up to Detect Diaphragm Injury and Herniation, in Patients With Asymptomatic Left Thoracoabdominal Stab Wounds: A Prospective Randomized Controlled Study
Brief Title: Laparoscopy Versus Clinical Follow up to Detect Diaphragm Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, PH NAVSARIA, Assoc Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: mlhgid004
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Diaphragm Injury
Keywords: Diaphragm injury; Herniation
MeSH Terms: conditions — Hernia | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Other): Laparoscopy on a group of randomly selected patients with left thoracoabdominal stab wounds to obtain the incidence of occult diaphragm injury
  Interventions: Procedure: Laparoscopy
- Control (Active Comparator): Assess the incidence and clinical outcome of delayed diaphragm visceral herniation in the study group.
  Interventions: Other: Clinical follow up

INTERVENTIONS:
Procedure: Laparoscopy — Treatment group will undergo a laparoscopy, with repair of the diaphragm if injury found
  Arms: Treatment
Other: Clinical follow up — Control group will undergo no treatment except suturing of wounds and drainage of the hemo-pneumothorax, if present. Then clinical follow up.
  Arms: Control

SUMMARY:
Title: A randomized prospective study comparing non operative management with laparoscopic treatment in patients with a diaphragm injury following left thoracoabdominal stab wounds.

Aim of the Study: The aim of this study is to access the clinical outcome of potential occult diaphragm injuries in a group of patients presenting at the Groote Schuur trauma centre with left sided thoracoabdominal stab wounds, if an expectant non operative management course is taken.

Objects of the Study: To obtain the above mentioned aim the study will undertake;

* to do laparoscopy on a group of randomly selected patients with left thoracoabdominal stab wounds to obtain the incidence of occult diaphragm injury.
* to assess the incidence and clinical outcome of delayed diaphragm visceral herniation in the study group.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable patients
* Patients with penetrating stab wounds bounded by
* Superiorly the 4th intercostal space
* Lateral the tip of the left scapula
* Inferior by the left costal margin
* Medially by the sternum
* Signed informed consent

Exclusion Criteria:

* Hemodynamically unstable patients
* Previous penetrating injury to the area mentioned under inclusion criteria
* Patients requiring early surgical exploration for injuries other than diaphragm injuries
* If a diaphragm injury is detected on imaging
* A positive pregnancy test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2009-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To assess the clinical outcome of potential occult diaphragm injuries in patients presenting at the Groote Schuur trauma centre with left sided thoracoabdominal stab wounds, if an expectant non operative management course is taken. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Navsaria, FCS (SA), Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa